CLINICAL TRIAL: NCT00659867
Title: Chromoscopy-guided Endomicroscopy With the PENTAX EC-3870CIFK / EC-3870CILK Confocal Colonoscopes for the Detection of Intraepithelial Neoplasias in Subjects With Long Standing Ulcerative Colitis
Brief Title: Endomicroscopy in Ulcerative Colitis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment problems
Sponsor: PENTAX Europe GmbH (Industry)
Collaborators: Johannes Gutenberg University Mainz (Other)
Responsible Party: Principal Investigator, Annette Weissmann, Trial Coordinator, PENTAX Europe GmbH
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 2006-09
Record Dates: First submitted 2008-04-14; First posted 2008-04-16 (Estimated); Last update posted 2016-09-27 (Estimated); Status verified 2016-09

CONDITIONS: Ulcerative Colitis
Keywords: Ulcerative Colitis; Endomicroscopy; Chromoendoscopy; Confocal colonoscope; Surveillance colonoscopy
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Chromoscopy-guided endomicroscopy with targeted biopsies
  Interventions: Device: PENTAX EC-3870CIFK / EC-3870CILK confocal colonoscopes
- B (Active Comparator): Standard endoscopy with random and targeted biopsies
  Interventions: Device: PENTAX EC-3870CIFK / EC-3870CILK confocal colonoscopes

INTERVENTIONS:
Device: PENTAX EC-3870CIFK / EC-3870CILK confocal colonoscopes — chromoscopy-guided endomicroscopy with targeted biopsies
  Other Names: Endomicroscope
  Arms: A
Device: PENTAX EC-3870CIFK / EC-3870CILK confocal colonoscopes — Standard endoscopy with random and targeted biopsies
  Other Names: Endomicroscope
  Arms: B

SUMMARY:
This is a confirmatory, multicentric, prospective, randomized, controlled, single-blind study in subjects with long standing ulcerative colitis in clinical remission with indication for surveillance colonoscopy. The patients are examined with the PENTAX EC-3870CIFK and EC-3870CILK confocal colonoscopes either by chromoscopy-guided endomicroscopy with targeted biopsies or by standard endoscopy with random and targeted biopsies. The aim is to investigate whether chromoscopy-guided endomicroscopy has a higher sensitivity than standard endoscopy with respect to detection of intraepithelial neoplasia (IN) and to compare the proportion of patients with at least 1 IN detected by chromoscopy-guided endomicroscopy versus standard endoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent must be available before any trial-related procedures
* Male and female patients aged 18 years and older
* Clinically and histologically verified UC
* Duration or Colitis ulcerosa >8 years (date of first diagnosis)
* Colitis Activity Index ≤ 8
* Activity index of Truelove and Witts: mild
* Ability of subject to understand character and individual consequences of clinical trial
* For women with childbearing potential, adequate contraception.

Exclusion Criteria:

* Known intraepithelial neoplasia or colorectal cancer
* Coagulopathy (Prothrombin time <50% of control, Partial thromboplastin time >50 s)
* Impaired renal function (Creatinine >1.2 mg/dL)
* Pregnancy or breast feeding
* Inability to obtain informed consent
* Active GI Bleeding
* Known allergy to methylene blue or fluorescein
* Participation in other clinical trials within the last 4 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Actual)
Dates: Start 2008-12; Primary Completion 2015-07 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
The primary objective is to investigate whether chromoscopy-guided endomicroscopy has a higher sensitivity than standard endoscopy with respect to detection of IN and to compare the proportion of patients with at least one IN | Day 1 (colonoscopy)

SECONDARY OUTCOMES:
Efficacy of chromoscopy-guided endomicroscopy in the detection of lesions and in the reduction of the number of biopsies. Time needed for the examination will be measured and compared between the two groups. | Day 1 (colonoscopy)

CONTACTS AND LOCATIONS:
Overall Officials: Ralf Kiesslich, Prof. Dr., Principal Investigator — Johannes Gutenberg-Universität Mainz, I. Med. Klinik
Locations (5):
- Germany (3):
  - Charité Campus Benjamin Franklin, Medizinische Klinik I, Berlin
  - Friedrich-Schiller-Universität Jena, Klinik für Innere Medizin II, Jena
  - Johannes Gutenberg-Universität Mainz, I. Med. Klinik und Poliklinik, Mainz
- Italy (2):
  - Ospedale Maggiore di Crema, Endoscopy and Gastroenterology Division, Crema
  - European Institute of Oncology, Division of Endoscopy, Milan

REFERENCES:
- [Background] Hurlstone DP, Kiesslich R, Thomson M, Atkinson R, Cross SS. Confocal chromoscopic endomicroscopy is superior to chromoscopy alone for the detection and characterisation of intraepithelial neoplasia in chronic ulcerative colitis. Gut. 2008 Feb;57(2):196-204. doi: 10.1136/gut.2007.131359. PMID 18192453 (Retraction: PMID 18949845 Gut. 2008 Nov;57(11):1634)